CLINICAL TRIAL: NCT03931122
Title: Comparison of Weight-based Versus External Ear-size Based Technique for Selection of Laryngeal Mask Airway in Pediatric Surgical Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Muhammad Qamarul Hoda, Professor, Department of Anesthesiology, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019-0246-3299
Record Dates: First submitted 2019-04-20; First posted 2019-04-30 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Laryngeal Masks; Minors; Child; Pediatrics
Keywords: Ear Size

STUDY DESIGN:
Intervention Model Description: All Laryngeal Mask Airways (LMA) devices being used in the study will be Ambu® AuraOnce™ (Ambu® A/S Baltorpbakken 13 DK-2750 Ballerup, Denmark) LMA's.
  LMA Size Selection: will be done for each patient according to group allocation:
  Group A - Weight based method Group B - Ear Size Based method
  Randomization technique:
  Patients will be randomized according to computer-generated blocked randomization (https://www.sealedenvelope.com) with blocks size of 6, by independent statistician (Anaesthesia research cell). Allocation concealment will be ensured by enclosing assignments in sealed, opaque, sequentially numbered envelopes which will be opened by one of the investigator only upon arrival of the patient in the operation room.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: One of the investigators will record patients' weight and external ear measurements in the study proforma. Patient's medical record (MR) number will then be send to the Research assistant/ Statistician for randomization into one of the groups (Group A or Group B). On the day of surgery, research assistant will hand over patient's group allocation in a sealed opaque envelop to one of the investigators who will not be the primary anesthetist. This investigator will determine the LMA size according to the group allocation. In case the dimensions fall between the two sizes of LMA in the ear size group, the closest one will be selected. After writing LMA size in the proforma it will be handed over to the primary anesthetist who will be blinded to patient's group allocation. Primary anesthetist (who has an experience of minimum 50 LMA insertions) will use the LMA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Weight Based Method (No Intervention): Body Weight Based method: This is the conventional method for LMA size selection. The patient will be weighed and LMA size corresponding to their weight will be used as follows.
  (LMA Size - 1 for up to 5 kg of body weight) (LMA Size - 1.5 for 5 to 10 kg of body weight) (LMA Size - 2 for 10 to 20 kg of body weight) (LMA Size - 2.5 for 20 to 30 kg of body weight) (LMA Size - 3 for 30 to 50 kg of body weight)
- Group B - Ear Size Based Method (Experimental): Ear Size Based method: External ear size will be measured by using a paper ruler and will be recorded in cm as follows:
  Vertical length: will be measured from the most dependent portion of the lobule to the furthest portion of the auricle.
  Horizontal length (width): from the tragus to the furthest part of the helix horizontally.
  Dimension(cm2): Vertical length (L) × Horizontal length (width-W )
  Based on these ear measurements, nearest smaller LMA size will be selected.
  Interventions: Device: Ear Size Based Method (Ambu® AuraOnce™ Laryngeal Mask Airway)

INTERVENTIONS:
Device: Ear Size Based Method (Ambu® AuraOnce™ Laryngeal Mask Airway) — The Laryngeal Mask Airway (LMA) is one of the devices used to maintain airway during general anesthesia. Its appropriate size is selected according to patients body weight as recommended by the manufacturer.
  However its appropriate size can also be selected via several other methods and one of them is patients external ear size. In this study the investigators will compare external ear size based method for LMA selection with the standard weight based method for LMA size selection.
  Vertical Ear length: will be measured from the most dependent portion of the lobule to the furthest portion of the auricle.
  Horizontal Ear length (width): from the tragus to the furthest part of the helix horizontally.
  Dimension(cm2): Vertical length (L) × Horizontal length (width-W)
  LMA Size LMA Cuff Length (cm) corresponding to vertical ear length.
  LMA Cuff Width (cm) corresponding to horizontal ear width.
  Arms: Group B - Ear Size Based Method

SUMMARY:
Laryngeal Mask Airway (LMA) is widely used in pediatric surgical patients. The manufacturer recommends the size of LMA to be used in children should be based on actual body weight but this method has several limitations. To overcome these concerns, various alternatives have been tried by different researchers, one of them is external ear size for LMA size selection. Investigators therefore would like to know whether the external ear size based method can be used for LMA size selection in pediatric surgical patients in Pakistan.

DETAILED DESCRIPTION:
OBJECTIVE:

to determine whether external ear-size is non-inferior to weight for LMA size selection in pediatric surgical patients.

INTRODUCTION:

The Laryngeal Mask Airway (LMA) is widely used in pediatric population. The manufacturer recommends the size of LMA to be used in children should be based on actual body weight. However, this method has several limitations, the range of weight for a particular size is very wide, it may not be appropriate for overweight or underweight children as it is based on actual body weight rather than ideal body weight, in emergency situations where weight of the patient is unknown the correlation between weight and size of LMA is impossible, and finally weight based recommendation may not be suitable as development of the child's oropharyngeal cavity is related to height and age rather than weight. All these factors may lead to inappropriate size selection, which may result in larger sized LMA causing trauma/injury to the airway and smaller ones causing obstruction or insufficient ventilation. To overcome these concerns various alternatives to weight based technique have been tried by different researchers in both adult and pediatric patients, one of them is external ear size. Literature revealed differences in external ear size dimensions in different ethnic population and the investigator's literature search failed to reveal any local data/study in Pakistani pediatric patients where external ear size was compared or used for size selection of the LMA. The investigators therefore would like to know whether the external ear size based method can be used for LMA size selection in pediatric surgical patients in Pakistan.

HYPOTHESIS:

External ear-size based technique is not inferior to weight based technique for LMA selection in pediatric population.

ELIGIBILITY:
Inclusion Criteria:

1. All children aged between 6 months to 18 years of age of either sex
2. American Society of Anesthesiologist (ASA) Classification I-II
3. Elective surgical procedures in whom an LMA will be indicated
4. Procedure lasting up to 2hrs

Exclusion Criteria:

1. Any external ear morphological abnormality
2. Previous external ear surgeries
3. Patient/Parent refusal
4. Children with oropharyngeal lesion
5. Any patient conditions (Gastroesophageal Re-flux Disease [GERD], hiatal hernia, incomplete NPO, bowel obstruction etc.) or procedures requiring rapid sequence induction and intubation
6. History of Upper respiratory tract infection (URTI) within the last 2 weeks

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 136 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Proper Placement | 1 minute
  Proper LMA placement will be assessed by chest expansion on positive pressure ventilation, absence of audible leak and a square wave capnograph waveform.
Adequacy of Ventilation | 1 minute
  Adequacy of ventilation: will be judged by an oxygen saturation of greater than or equal to 95% at a Fractional Inspired Oxygen concentration (FiO2) less than 0.5 and an end-tidal carbon dioxide (ETCO2) of 35-45 mmHg at a tidal volume of 6- 8 ml/kg Actual Body Weight (ABW) at peak airway pressure less than the oropharyngeal leak pressure (OLP), and by adjusting the respiratory rate (RR).

SECONDARY OUTCOMES:
Oropharyngeal Leak Pressure (OLP) | 30 seconds
  Oropharyngeal Leak Pressure (OLP): will be determined at LMA intra-cuff pressure of 60 cmH2O by closing the Adjustable Pressure Limiting (APL) valve of the circle system at a fixed gas flow of 3 Liters per minute and by noting the circuit pressure at which an equilibrium will be reached and then releasing it completely.
Leak fraction (LF) | 1 minute
  Leak fraction (LF): will be determined by comparing the difference between inspired and expired tidal volumes and dividing them by the inspired tidal volume at a tidal volume (TV) of 8 ml/kg actual body weight (ABW) with an I:E ratio of 1:2 and respiratory rate (RR) of 20 breaths per minute.
Incidence of mucosal injury and laryngospasm | 1 minute
  Incidence of mucosal injury in the two groups will be assessed by trauma or minor injury to the airway seen as blood on the device after removal.
  Incidence of laryngospasm will also be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Qamarul Hoda, FCAI, Principal Investigator — The Aga Khan University Hospital, Karachi, Pakistan.; Muhammad Asghar Ali, FCPS, Principal Investigator — The Aga Khan University Hospital, Karachi, Pakistan.; Hameed Ullah, FCPS, Principal Investigator — The Aga Khan University Hospital, Karachi, Pakistan.; Samie Asghar Dogar, FCPS, Principal Investigator — The Aga Khan University Hospital, Karachi, Pakistan.; Muhammad Saad Yousuf, FCPS, Principal Investigator — The Aga Khan University Hospital, Karachi, Pakistan.; Bushra Salim, FCPS, Principal Investigator — The Aga Khan University Hospital, Karachi, Pakistan.
Locations (1):
- Muhammad Asghar Ali, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The investigators will not publish any identifiable data, it will remain confidential. However the investigators will present this study in local and international meetings and also publish it in local or international journal.
Supporting Information: CSR
Time Frame: The data would be handled by the primary investigator and hard copies of the data will be saved by a lock and key method and soft copies will be saved on a computer and the data will be password protected. It will become available 6 months after completion of the study. Due to a regulatory requirement, this data will be saved for 15 years.

REFERENCES:
- [Background] Lopez-Gil M, Brimacombe J, Alvarez M. Safety and efficacy of the laryngeal mask airway. A prospective survey of 1400 children. Anaesthesia. 1996 Oct;51(10):969-72. doi: 10.1111/j.1365-2044.1996.tb14968.x. PMID 8984875
- [Background] Kim MS, Lee JS, Nam SB, Kang HJ, Kim JE. Randomized Comparison of Actual and Ideal Body Weight for Size Selection of the Laryngeal Mask Airway Classic in Overweight Patients. J Korean Med Sci. 2015 Aug;30(8):1197-202. doi: 10.3346/jkms.2015.30.8.1197. Epub 2015 Jul 15. PMID 26240500
- [Background] Kim HJ, Park MJ, Kim JT, Kim CS, Kim SD, Kim HS. Appropriate laryngeal mask airway size for overweight and underweight children. Anaesthesia. 2010 Jan;65(1):50-3. doi: 10.1111/j.1365-2044.2009.06160.x. Epub 2009 Nov 17. PMID 19922510
- [Background] Ho AM, Karmakar MK, Dion PW. Choosing the correct laryngeal mask airway sizes and cuff inflation volumes in pediatric patients. J Emerg Med. 2008 Oct;35(3):299-300. doi: 10.1016/j.jemermed.2007.10.073. Epub 2008 May 7. PMID 18462912
- [Background] Rommel N, Bellon E, Hermans R, Smet M, De Meyer AM, Feenstra L, Dejaeger E, Veereman-Wauters G. Development of the orohypopharyngeal cavity in normal infants and young children. Cleft Palate Craniofac J. 2003 Nov;40(6):606-11. doi: 10.1597/1545-1569_2003_040_0606_dotoci_2.0.co_2. PMID 14577816
- [Background] Tang MY, Tang IP, Wang CY. Optimal Size AMBU(R) Laryngeal Mask Airway Among Asian Adult Population. Med J Malaysia. 2014 Aug;69(4):151-5. PMID 25500841
- [Background] Devitt JH, Wenstone R, Noel AG, O'Donnell MP. The laryngeal mask airway and positive-pressure ventilation. Anesthesiology. 1994 Mar;80(3):550-5. doi: 10.1097/00000542-199403000-00011. PMID 8141451
- [Background] Huang YH, Cherng CH. Optimal size selection of the classic laryngeal mask airway by tongue width-based method in male adults. J Chin Med Assoc. 2014 Aug;77(8):422-5. doi: 10.1016/j.jcma.2014.05.009. Epub 2014 Jul 16. PMID 25043385
- [Background] Weng M, Ding M, Xu Y, Yang X, Li L, Zhong J, Miao C. An Evaluation of Thyromental Distance-based Method or Weight-based Method in Determining the Size of the Laryngeal Mask Airway Supreme: A Randomized Controlled Study. Medicine (Baltimore). 2016 Mar;95(9):e2902. doi: 10.1097/MD.0000000000002902. PMID 26945383
- [Background] Gallart L, Mases A, Martinez J, Montes A, Fernandez-Galinski S, Puig MM. Simple method to determine the size of the laryngeal mask airway in children. Eur J Anaesthesiol. 2003 Jul;20(7):570-4. doi: 10.1017/s0265021503000917. PMID 12884992
- [Background] Zahoor A, Ahmad N, Sereche G, Riad W. A novel method for laryngeal mask airway size selection in paediatric patients. Eur J Anaesthesiol. 2012 Aug;29(8):386-90. doi: 10.1097/EJA.0b013e32835562f4. PMID 22692042
- [Background] Haliloglu M, Bilgen S, Uzture N, Koner O. [Simple method for determining the size of the ProSeal laryngeal mask airway in children: a prospective observational study]. Rev Bras Anestesiol. 2017 Jan-Feb;67(1):15-20. doi: 10.1016/j.bjan.2016.09.007. Epub 2016 Sep 29. Portuguese. PMID 27692804
- [Background] Alexander KS, Stott DJ, Sivakumar B, Kang N. A morphometric study of the human ear. J Plast Reconstr Aesthet Surg. 2011 Jan;64(1):41-7. doi: 10.1016/j.bjps.2010.04.005. Epub 2010 May 5. PMID 20447883
- [Background] Suzanna AB, Liu CY, Rozaidi SW, Ooi JS. Comparison between LMA-Classic and AMBU AuraOnce laryngeal mask airway in patients undergoing elective general anaesthesia with positive pressure ventilation. Med J Malaysia. 2011 Oct;66(4):304-7. PMID 22299547
- [Background] Jagannathan N, Hajduk J, Sohn L, Huang A, Sawardekar A, Gebhardt ER, Johnson K, De Oliveira GS. A randomised comparison of the Ambu(R) AuraGain and the LMA(R) supreme in infants and children. Anaesthesia. 2016 Feb;71(2):205-12. doi: 10.1111/anae.13330. Epub 2015 Dec 9. PMID 26648173
- [Background] Natalini G, Franceschetti ME, Pantelidi MT, Rosano A, Lanza G, Bernardini A. Comparison of the standard laryngeal mask airway and the ProSeal laryngeal mask airway in obese patients. Br J Anaesth. 2003 Mar;90(3):323-6. doi: 10.1093/bja/aeg060. PMID 12594145
- [Background] Bordes M, Semjen F, Degryse C, Bourgain JL, Cros AM. Pressure-controlled ventilation is superior to volume-controlled ventilation with a laryngeal mask airway in children. Acta Anaesthesiol Scand. 2007 Jan;51(1):82-5. doi: 10.1111/j.1399-6576.2006.01148.x. Epub 2006 Nov 1. PMID 17073863
- [Background] Park C, Bahk JH, Ahn WS, Do SH, Lee KH. The laryngeal mask airway in infants and children. Can J Anaesth. 2001 Apr;48(4):413-7. doi: 10.1007/BF03014975. PMID 11339788
- [Background] von Ungern-Sternberg BS, Boda K, Schwab C, Sims C, Johnson C, Habre W. Laryngeal mask airway is associated with an increased incidence of adverse respiratory events in children with recent upper respiratory tract infections. Anesthesiology. 2007 Nov;107(5):714-9. doi: 10.1097/01.anes.0000286925.25272.b5. PMID 18073545
- [Background] Hemmerling TM, Beaulieu P, Jacobi KE, Babin D, Schmidt J. Neuromuscular blockade does not change the incidence or severity of pharyngolaryngeal discomfort after LMA anesthesia. Can J Anaesth. 2004 Aug-Sep;51(7):728-32. doi: 10.1007/BF03018434. PMID 15310644
- [Background] Das B, Mitra S, Samanta A, Samal RK. A comparative study of three methods of ProSeal laryngeal mask airway insertion in children with simulated difficult laryngoscopy using a rigid neck collar. Acta Anaesthesiol Taiwan. 2014 Sep;52(3):110-3. doi: 10.1016/j.aat.2014.05.009. Epub 2014 Jul 26. PMID 25073752
- [Background] Adamus M, Belohlavek R, Koutna J, Vujcikova M, Janaskova E. Cisatracurium vs. Rocuronium: A prospective, comparative, randomized study in adult patients under total intravenous anaesthesia. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2006 Nov;150(2):333-8. doi: 10.5507/bp.2006.051. PMID 17426802
- [Background] El-Boghdadly K, Bailey CR, Wiles MD. Postoperative sore throat: a systematic review. Anaesthesia. 2016 Jun;71(6):706-17. doi: 10.1111/anae.13438. Epub 2016 Mar 28. PMID 27158989
- [Background] Al-Sunduqchi MS. Determining the Appropriate Sample Size for Inferences Based on the Wilcoxon Statistics. Ph.D. dissertation under the direction of William C. Guenther, Dept. of Statistics, University of Wyoming, Laramie, Wyoming. 1990.
- [Background] Chow S-C, Shao J WH. Sample Size Calculations in Clinical Research. New York.: Marcel Dekker.; 2003.
- [Background] Julious SA. Sample sizes for clinical trials with normal data. Stat Med. 2004 Jun 30;23(12):1921-86. doi: 10.1002/sim.1783. PMID 15195324
- [Background] Meretoja OA, Taivainen T, Wirtavuori K. Pharmacodynamic effects of 51W89, an isomer of atracurium, in children during halothane anaesthesia. Br J Anaesth. 1995 Jan;74(1):6-11. doi: 10.1093/bja/74.1.6. PMID 7880708
- [Background] Fuchs-Buder T, Baumann C, De Guis J, Guerci P, Meistelman C. Low-dose neostigmine to antagonise shallow atracurium neuromuscular block during inhalational anaesthesia: A randomised controlled trial. Eur J Anaesthesiol. 2013 Oct;30(10):594-8. doi: 10.1097/EJA.0b013e3283631652. PMID 23803594